CLINICAL TRIAL: NCT05895461
Title: Developing a Behavioral Weight Loss Intervention for Emerging Adults Implemented Within College Health Service Centers
Brief Title: Weight Management Intervention in College: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1793732; K23DK128561 (NIH)
Record Dates: First submitted 2023-05-22; First posted 2023-06-08 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2024-09

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity

STUDY DESIGN:
Intervention Model Description: The first 3 cohorts of this study were a single group pre-post design. Based on findings from those, the fourth cohort was changed to include a control group (arm 2). A control group was not originally planned until the next phase of the study; however, it was included at this stage in order to put achievement of weight benchmarks into context and inform potential progression decision-making.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- BWLI-College (Experimental): BWLI-College is a multicomponent behavioral weight loss intervention to reduce weight through diet, physical activity, and behavioral modifications designed to be responsive to emerging adult preferences. It will be delivered in a hybrid format with in-person and remotely-delivered asynchronous sessions. As presently designed, the intervention will last 10 weeks, though this may change with refinement.
  Interventions: Behavioral: BWLI-College
- Control (Active Comparator): The Control intervention consists of 1 in-person psychoeducational group session on general weight loss information and myths. Public web-resources about healthy eating and physical activity will be provided. Newsletters with similar content will be sent to promote retention.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: BWLI-College — Behavioral modifications are based on empirically-supported principles for weight loss.
  Diet recommendations follow a small change approach in which participants will make a series of small, self-selected dietary changes each day (~100-200 calories) that they build on over the course of the intervention.
  Physical activity recommendations are to achieve 150-250 weekly minutes of moderate-to-vigorous physical activity with specific goals and rate of progression that are individualized to each participant.
  Arms: BWLI-College
Behavioral: Control — Psychoeducation around dieting myths, healthy eating, and physical activity
  Arms: Control

SUMMARY:
This Proof-of-Concept study consists of a series of uncontrolled pilot studies to refine a behavioral weight loss trial using a "small change" approach for emerging adult college students with overweight/obesity. The primary aim of this study is maximize student acceptability of the intervention and weight loss outcomes.

DETAILED DESCRIPTION:
Forty percent of emerging adults (age 18-25) have overweight or obesity, which is unlikely to remit and has significant health consequences. However, emerging adults are underrepresented in traditional weight loss programs, drop-out at high rates, and have blunted weight loss outcomes. One potential way to improve participation is to offer BWLIs in college health service centers to reduce barriers to participation. Approximately 40% of emerging adults are enrolled in a postsecondary institution and college health centers are used widely by students. Moreover, delivering an intervention with design features that are responsive to emerging adult preferences and lifestyles may also improve intervention effectiveness and attractiveness. The "small change" (SC) approach to weight loss addresses emerging adult barriers to engagement by focusing on reducing calories through a few self-selected, specific changes to current obesogenic behaviors, requiring less time and effort than traditional behavioral weight loss interventions (BWLI) and promoting autonomy and self-efficacy. The SC approach has been used effectively for weight loss in other populations. This proof-of-concept study is part of a larger study that aims to develop and refine a novel and effective BWLI based on a SC approach that is designed for emerging adults and for implementation in college health centers, an accessible care setting. The primary aim of this proof-of-concept study is to iteratively test and refine the intervention to maximize student acceptability and weight loss outcomes.

ELIGIBILITY:
Inclusion Criteria:

* BMI of 25 or greater
* Enrolled at college/university where study will take place
* English-speaking

Exclusion Criteria:

* History or current diagnosis of anorexia nervosa, bulimia nervosa, or alcohol use disorder (current symptoms also assessed at screening using validated screening questionnaires)
* Participation in another formal weight loss program
* Current or recent pregnancy
* Psychiatric hospitalization in the past 12 months
* Recent weight loss of 5% body weight or more
* History of bariatric surgery
* Severe food or physical activity restrictions that would interfere with treatment recommendations

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2023-05-08 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline F Hayes, PhD, Principal Investigator — Brown University
Locations (1):
- The Miriam Hospital, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be made available to share with other researchers.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment in this trial followed college semesters, starting in Summer 2023 and ending in Fall 2024.
Pre-assignment Details: While 42 signed the consent, n=6 were unable to participate due to their scheduling (i.e., their schedule did not allow for them to participate at the selected time) and n=2 were lost to follow-up prior to initiating treatment and learning of treatment condition.
Groups:
- BWLI-College: BWLI-College is a multicomponent behavioral weight loss intervention to reduce weight through diet, physical activity, and behavioral modifications designed to be responsive to emerging adult preferences. It will be delivered in a hybrid format with in-person and remotely-delivered asynchronous sessions. As presently designed, the intervention will last 10 weeks, though this may change with refinement.
  BWLI-College: Behavioral modifications are based on empirically-supported principles for weight loss.
  Diet recommendations follow a small change approach in which participants will make a series of small, self-selected dietary changes each day (~100-200 calories) that they build on over the course of the intervention.
  Physical activity recommendations are to achieve 150-250 weekly minutes of moderate-to-vigorous physical activity with specific goals and rate of progression that are individualized to each participant.
Period: Overall Study
Arm/Group | BWLI-College | Control
Started | 29 | 5
Completed | 24 | 5
Not Completed | 5 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | BWLI-College | Control | Total
Number analyzed (Participants) | 29 | 5 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 29 | 5 | 34
  >=65 years | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 5 | 0 | 5
  White | 19 | 3 | 22
  More than one race | 2 | 1 | 3
  Unknown or Not Reported | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 8 | 2 | 10
  Not Hispanic or Latino | 21 | 3 | 24
  Unknown or Not Reported | 0 | 0 | 0
Weight Category [Count of Participants; unit: Participants]
  Overweight | 6 | 1 | 7
  Obese | 23 | 4 | 27
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 3 | 29
  Male | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Acceptability
Description: Refers to the satisfactory nature of a treatment and will be assessed via the 4-item Acceptability of Intervention Measure. Benchmarks are to reach mean scores of at least 4 out of 5. Range is 1 to 5, with higher scores indicating greater acceptability.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: score
Arm/Group | BWLI-College | Control
Number analyzed (Participants) | 24 | 5
score | 4.6 (0.5) | 4.2 (0.8)

2. Primary Outcome: Percentage of Participants Who Remained at 10 Weeks
Description: Rate of retention of 80% or more (benchmark)
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | BWLI-College | Control
Number analyzed (Participants) | 29 | 5
Participants | 24 | 5

3. Primary Outcome: Adherence
Description: Average attendance and completion of sessions of 75% or more (benchmark)
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: percent sessions attended
Arm/Group | BWLI-College | Control
Number analyzed (Participants) | 24 | 5
percent sessions attended | 77.5 (20.2) | 80 (44.7)

4. Primary Outcome: Weight Change
Description: Average weight loss of at least 3% (benchmark)
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | BWLI-College | Control
Number analyzed (Participants) | 24 | 5
percent change | -1.7 (2.8) | 0.7 (3.4)

ADVERSE EVENTS:
Time Frame: from enrollment until end of follow-up, up to 10 weeks
Description: Collection approach was non-systematic for initial cohorts and a questionnaire (systematic) process was added.
Arm/Group | BWLI-College | Control
All-Cause Mortality (participants affected / at risk) | 0/29 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/29 | 0/5
Other Adverse Events (participants affected / at risk) | 3/29 | 2/5
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | BWLI-College (N=29) | Control (N=5)
Treatment initiation or change (Psychiatric disorders) | 3 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-08-19): https://cdn.clinicaltrials.gov/large-docs/61/NCT05895461/Prot_SAP_000.pdf